CLINICAL TRIAL: NCT02083445
Title: Exercise, Muscle Electro-stimulation and Intermittent Hypobaric Hypoxia Program and Circulating Progenitor Cells in Traumatic Brain Injured Patients
Brief Title: Exercise, Hypoxia and CPC in TBI Patients
Acronym: TCECAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Luisa Corral, Luisa Corral, University of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DEP2010-222005-C02-02; AC048-10, PR017/10 (Other: Comité de Ética de Investigación Clínica de Bellvitge)
Record Dates: First submitted 2014-03-01; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Exercise; Psychology; Physiology; Progenitor cells; Hypoxia
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity; Hypoxia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Placebo Comparator): Once a week there will be an attendance cognitive session (specific sessions designed to work on aspects related to body perception, movement, space) and the extraction of blood samples will be carried out to determine the progenitor cells on the same day of the active groups.
  Interventions: Other: cognitive activities
- Exercise group (Active Comparator): Patients with past history of TBI will perform exercise sessions two hours three days a week during 12 weeks. The sessions will consist of aerobic, strength, flexibility, proprioception and balance activities and muscle electro-stimulation sessions or cycling sessions.
  Interventions: Other: Exercise program
- Muscle electro-stimulation and IHH (Active Comparator): Patients with past history of TBI will perform a 12 weeks program: intermittent hypobaric hypoxia (IHH) 2 hours at a simulated altitude of 4500 meters 3 days/week. Muscle electro-stimulation for two periods of 20 minutes during the stay in the hypobaric chamber.
  Interventions: Device: Muscle electro-stimulation; Other: Intermittent hypobaric hypoxia

INTERVENTIONS:
Other: cognitive activities — Participants followed a day of cognitive activities 1 day (1 hour/day) per week during 12 weeks.
  Arms: Control group
Other: Exercise program — Exercise program of endurance, resistance and proprioception exercises, comprising three sessions per week and muscle electro-stimulation was applied using the Compex Vitality® vascular and capillarization program with electrodes fixed in quadriceps and abdominal muscles or cycling exercise.
  Arms: Exercise group
Device: Muscle electro-stimulation — A program of intermittent hypobaric hypoxia and muscle electro-stimulation of 3 days (3 hours/day) per week during 12 weeks
  Arms: Muscle electro-stimulation and IHH
Other: Intermittent hypobaric hypoxia
  Arms: Muscle electro-stimulation and IHH

SUMMARY:
Circulating progenitor cells (CPC) treatments may have great potential for the recovery of neurons and brain function. Our group has reported how exposure to intermittent hypobaric hypoxia with superficial muscle electrostimulation is able to increase the concentration of CPC in peripheral blood in humans. Therefore, we believe that through physical activities and exposure to intermittent hypobaric hypoxia for a period, it will increase CPC in the blood of subjects who have suffered a severe Traumatic Brain Injury (TBI) one or more years ago, promoting regeneration and functional and cognitive recovery. The study primary end-point is to improve physical or psychological functioning of participants with TBI with a program of exercise, muscle electro-stimulation (ME) and/or intermittent-hypobaric-hypoxia (IHH). Secondary end-points are to increase and maintain CPC and also to study their possible relationship with physical or psychological improvement of participants with Traumatic Brain Injury (TBI). In order to achieve these objectives investigators have designed a randomized controlled trial that will include those patients who suffered severe TBI more than one year previously with physical or psychological sequelae. Exercise, muscle electro-stimulation (ME) and/or intermittent hypobaric hypoxia (IHH) programs will be applied during twelve weeks. Psychological and physical stress tests will carry out before and after the program and CPC will measure at the beginning, every two weeks, and at the end of the program.

DETAILED DESCRIPTION:
Clinical, experimental, case control and prospective study. Inclusion criteria are: patients who suffered severe TBI more than one year previously with physical or psychological sequelae, male sex, and age 20-60 years old. Patients with epilepsy are not included. The study was approved by the institution's Research Ethics Committee and informed consent was obtained from the patients.

A program of three days per week during twelve weeks will be applied to the active groups: one, exercise and muscle electrical stimulation, and the other, exercise, muscle electrical stimulation and IHH chamber exposure. Control group participants will follow a a day of cognitive activities one day per week during 12 weeks.

Psychological and physical stress tests are carried out before and after the program. Psychological tests evaluate features of language and work (verbal memory-RAVLT), Trail Making Test (TMT A and B), Stroop Test, working memory capacity and attention (WAIS III), information processing speed (WAIS III), orientation and verbal fluency (Barcelona test), executive functions (WAIS III and Tower of London tests) and estimated premorbid intelligence index (vocabulary, WAIS III). Reduced Paced Auditory Serial Addition Test (PASAT-G) evaluate work memory components. Physical graded maximum stress tests were performed on a cycle ergometer increasing progressively the workload, in order to evaluate physical capacity and adaptation to different intensities of effort. CPC (CD34+) are measured in peripheral blood according to a previously used method (Viscor et al., 2009), at the beginning, every two weeks, and at the end of the program (blood samples were always obtained before the exercise sessions).

Statistical analysis: data will express as mean, median, standard deviation and interquartile range as appropriate. The continuous variables will compare using the Mann-Whitney U test. Wilcoxon signed rank test and Friedman test are used for repeated measures. All tests will perform using Statistical Package for the Social Sciences (SPSS) v.13. Statistical significance was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffered severe TBI more than one year previously with physical or psychological sequelae.
* Written informed consent from patient

Exclusion Criteria:

* Epilepsy
* Any medical or psychological contraindications for implementing the program of physical activity or hypobaric chamber.
* Inclusion in other ongoing study
* Refuse consent

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from initial physical stress test at one week post-intervention | One week before and an expected average of one week after the intervention
  Physical graded maximum stress tests are performed on a cycle ergometer controlling the workload, in order to evaluate physical capacity and adaptation to different intensities of effort.While performance of these tests are conducted, cardiocirculatory (control of heart rate, blood pressure measurement, continuous ECG) and respiratory (breathing gases analysis) are monitored to observe the adaptation to the effort.
Change from initial psychological test at one weeks after intervention | One week before and an average of one week after the intervention
  Psychological tests evaluated features of language and work (verbal memory-RAVLT), Trail Making Test (TMT A and B), Stroop Test, working memory capacity and attention (WAIS III), information processing speed (WAIS III), orientation and verbal fluency (Barcelona test), executive functions (WAIS III and Tower of London tests) and estimated premorbid intelligence index (vocabulary, WAIS III). Reduced Paced Auditory Serial Addition Test (PASAT-G)

SECONDARY OUTCOMES:
Circulating progenitor cells increase | The day before, every 15 days during the intervention and two weeks after the intervention
  Blood CD34 staining and flow cytometry assay in accordance with ISHAGE guidelines (Keeney et al., 1998). CD34 cells/µL.

OTHER OUTCOMES:
Relationship between circulating progenitor cells and physical or psychological tests improvement | An average of two weeks after intervention
  If a statistically significant increase of circulating progenitor cells occurs and physical and/or psychological tests improvement, their relationship will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Corral, MD, PhD, Principal Investigator — University of Barcelona and Bellvitge University Hospital; Casimiro F Javierre, MD, PhD, Study Director — Universiy of Barcelona; Ginés Viscor, PhD, Study Chair — University of Barcelona; Josep L Ventura, MD, PhD, Study Director — Bellvitge University Hospital
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Viscor G, Javierre C, Pages T, Ventura JL, Ricart A, Martin-Henao G, Azqueta C, Segura R. Combined intermittent hypoxia and surface muscle electrostimulation as a method to increase peripheral blood progenitor cell concentration. J Transl Med. 2009 Oct 29;7:91. doi: 10.1186/1479-5876-7-91. PMID 19874615
- [Background] Corral L, Javierre CF, Ventura JL, Marcos P, Herrero JI, Manez R. Impact of non-neurological complications in severe traumatic brain injury outcome. Crit Care. 2012 Dec 12;16(2):R44. doi: 10.1186/cc11243. PMID 22410278
- [Background] Corral L, Ventura JL, Herrero JI, Monfort JL, Juncadella M, Gabarros A, Bartolome C, Javierre CF, Garcia-Huete L. Improvement in GOS and GOSE scores 6 and 12 months after severe traumatic brain injury. Brain Inj. 2007 Nov;21(12):1225-31. doi: 10.1080/02699050701727460. PMID 18236198
- [Background] Bennie SD, Petrofsky JS, Nisperos J, Tsurudome M, Laymon M. Toward the optimal waveform for electrical stimulation of human muscle. Eur J Appl Physiol. 2002 Nov;88(1-2):13-9. doi: 10.1007/s00421-002-0711-4. Epub 2002 Sep 10. PMID 12436266
- [Background] Bonsignore MR, Morici G, Riccioni R, Huertas A, Petrucci E, Veca M, Mariani G, Bonanno A, Chimenti L, Gioia M, Palange P, Testa U. Hemopoietic and angiogenetic progenitors in healthy athletes: different responses to endurance and maximal exercise. J Appl Physiol (1985). 2010 Jul;109(1):60-7. doi: 10.1152/japplphysiol.01344.2009. Epub 2010 May 6. PMID 20448032
- [Background] Driver S, Ede A. Impact of physical activity on mood after TBI. Brain Inj. 2009 Mar;23(3):203-12. doi: 10.1080/02699050802695574. PMID 19205956
- [Background] Guo X, Liu L, Zhang M, Bergeron A, Cui Z, Dong JF, Zhang J. Correlation of CD34+ cells with tissue angiogenesis after traumatic brain injury in a rat model. J Neurotrauma. 2009 Aug;26(8):1337-44. doi: 10.1089/neu.2008.0733. PMID 19226208
- [Background] Koutroumpi M, Dimopoulos S, Psarra K, Kyprianou T, Nanas S. Circulating endothelial and progenitor cells: Evidence from acute and long-term exercise effects. World J Cardiol. 2012 Dec 26;4(12):312-26. doi: 10.4330/wjc.v4.i12.312. PMID 23272272
- [Background] Ploughman M. Exercise is brain food: the effects of physical activity on cognitive function. Dev Neurorehabil. 2008 Jul;11(3):236-40. doi: 10.1080/17518420801997007. PMID 18781504
- [Background] Mobius-Winkler S, Hilberg T, Menzel K, Golla E, Burman A, Schuler G, Adams V. Time-dependent mobilization of circulating progenitor cells during strenuous exercise in healthy individuals. J Appl Physiol (1985). 2009 Dec;107(6):1943-50. doi: 10.1152/japplphysiol.00532.2009. Epub 2009 Oct 1. PMID 19797690
- [Background] Wang JS, Lee MY, Lien HY, Weng TP. Hypoxic exercise training improves cardiac/muscular hemodynamics and is associated with modulated circulating progenitor cells in sedentary men. Int J Cardiol. 2014 Jan 1;170(3):315-23. doi: 10.1016/j.ijcard.2013.11.005. Epub 2013 Nov 12. PMID 24286591
- [Background] Xu Q, Wang S, Jiang X, Zhao Y, Gao M, Zhang Y, Wang X, Tano K, Kanehara M, Zhang W, Ishida T. Hypoxia-induced astrocytes promote the migration of neural progenitor cells via vascular endothelial factor, stem cell factor, stromal-derived factor-1alpha and monocyte chemoattractant protein-1 upregulation in vitro. Clin Exp Pharmacol Physiol. 2007 Jul;34(7):624-31. doi: 10.1111/j.1440-1681.2007.04619.x. PMID 17581219
- [Background] Zhu LL, Zhao T, Li HS, Zhao H, Wu LY, Ding AS, Fan WH, Fan M. Neurogenesis in the adult rat brain after intermittent hypoxia. Brain Res. 2005 Sep 7;1055(1-2):1-6. doi: 10.1016/j.brainres.2005.04.075. PMID 16098951